CLINICAL TRIAL: NCT07155148
Title: Argentine Registry of Crohn's Disease and Ulcerative Colitis
Acronym: RADECCU
Status: Recruiting | Type: Observational
Sponsor: Grupo Argentino de Enfermedad de Crohn y Colitis Ulcerosa (Other)
Responsible Party: Sponsor
Other Study IDs: RADECCU
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Epidemiology; Inflammatory Bowel Disease (IBD); Therapy
Keywords: Crohn's Disease; Ulcerative Colitis; Argentina; Registry; Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study — Observational registry without clinical interventions

SUMMARY:
RADECCU is a strictly observational IBD registry in Argentina. The registry is open to all practicing gastroenterologist in the country grouped within the Argentinean Crohn's and Ulcerative Colitis Group (GADECCU). The registry will include outcomes of routine clinical practice of patients with IBD including the pediatric and adult population.

DETAILED DESCRIPTION:
Aims:

The primary objective of the registry is to create an IBD physicians' network in Argentina that captures pragmatic and relevant information from IBD patients in terms of demographic, clinical and diagnostic aspects. The secondary objective includes safety aspects, including infections, and access to healthcare. The tertiary objective is related to treatment effectiveness. For the treatment effectiveness outcome, information about IBD complications as flares, need of hospitalization and surgery will be included.

Structure of the registry:

The administrative structure of the registry includes an executive committee with an administrative and organizational role which is coordinating with the GADECCU steering committee; a scientific committee that evaluates and coordinates scientific initiatives and promotes specific new strategic projects of interest and approves requests for access to centralized data for research projects. Also, a methodological and regulatory team that provides methodological support to the registry and ensures the regulatory aspects in each institution or region. RADECCU includes a group of technical programmers who develop and provide support to the web platform that allows researchers to register and follow their patients.

Ethical aspects:

The RADECCU registry was approved by the ethics committee of each participant center with a similar project model. Later, individual regulatory and data protection requirements were fulfilled according to all applicable local regulations and laws in each participant center and practice. According the requirements of local approval of each center (need for informed consent or not) the principal investigator or those delegated to the center as co-investigators will fully explains the objective of the registry to all potential participants and encourages their questions. All patients willing to participate in the registry are required to provide an oral or signed consent form (pending on each approval) authorizing release of their coded medical information anonymized to the central registry. To be included in the registry, every center must fulfill the ethical and regulatory conditions.

Population:

Any patient diagnosed with IBD defined by validated diagnostic criteria can be included into the registry. The criteria for IBD diagnosis were agreed with all the members of the Scientific Committee of the registry prior to the start of registration, and were based on previously published criteria for IBD diagnosis, including clinical, endoscopic, laboratory, and histopathological aspects, as well as small bowel imaging studies (Bernstein CN, et al. Inflamm Bowel Dis. 2010;16(1):112-24. doi: 10.1002/ibd.21048.). In order to ensure the inclusion of all IBD patients in Argentina, the executive committee invites all centers associated to GADECCU and involved in the management of IBD patients, regardless of the volume of patients they are in charge of, including both public and private centers. To reduce the possibility of selection bias, each participating physician from each center should aim to include all patients seen in their practice or clinic.

Centers and physicians involved:

Medical assistance to IBD patients in Argentina is mainly provided by several physicians in different institutions and IBD unit throughout the country. The goal of the registry is to include all IBD patients in Argentina and, consequently, all IBD centers and physicians involved in the care of affected patients. All physicians and centers that are part of GADECCU were invited to participate in the registry. In addition, an invitation campaign was carried out at local and national gastroenterology congresses and scientific meetings for physicians not yet linked to GADECCU so that they could get to know and participate in the registry through GADECCU.

The participation in RADECCU is voluntary for both the physicians and the patient. From February-2023 an active promotion of the registry was carried out, resulting in a final incorporation of 65 centers and 138 professionals distributed throughout Argentina.

Data collection and patient confidentiality:

Prevalent and incident cases are included in the Registry by each physician. Once the patient is identified, the requested data is included in a web platform specifically designed for the purpose of the registry. The data is uploaded by the principal investigators of each participating center. The Scientific Committee of RADECCU agree in a prior consensus, on a compulsory common minimum dataset consisting of selected information according to the principles of relevance to ensure the collection of enough data for the clinical characterization of a single patient.

RADECCU is a website with restricted access only to authorized users with a username and password assigned by the executive committee. Users can only view the identifying data of patients they have uploaded themselves, and those who can access the complete database will only have access to an anonymized version of it. The platform will provide data in a comprehensive manner with low cost of development.

During all registration processes, the protection of the patient's identity and data is observed in accordance with the legal regulations in force under the National Law of Protection of Personal Data from Argentina 25.326 (Habeas Data), in accordance with the international legislation on registration of diseases and protection of personal and private data, according to the 18th World Medical Assembly of Helsinki (1964), when applicable. The right to non-participation in the registry is always respected without this implying in any case any type of discrimination, differential treatment or mistreatment towards the patient.

The entire process regarding informed consent, patient evaluation, data entry, data sharing and other procedures of the registry were standardized in an operation procedure described in documents of the registry function, and is available to all researchers in the registry.

Data monitoring:

The structure of the registry was designed considering all the mandatory variables at the time of entry and during the follow-up to be full upload. In this way, data loss is ensured to be kept at a minimum. Data will be centrally monitored by the methodological team to guarantee a high level of quality for the information collected. Centers will be periodically contacted with ad hoc reports with queries on missing data, inconsistencies among variables collected and any duplicates for their resolution.

Research projects:

The mission of RADECCU is not limited to assuring quality healthcare for patients with IBD in Argentina but also to stimulate research projects that address high-priority issues in our region. The philosophy behind the registry takes to reflect the collaborative nature of the project and to encourage epidemiological research efforts in IBD in Argentina. Any researcher who is part of the RADECCU may propose a research project with local or national impact that will be evaluated by the Scientific Committee and, if relevant, will be approved for its development. The data contained in the registry will be used in the research project and, in this way, the performance of various epidemiological studies employing data from RADECCU will also be stimulated.

Statistical analysis plan:

This is an open-ended registry, and sample size is not based on statistical considerations. The main objective of the Registry is a descriptive analysis regarding demographic and clinical aspects, therapy, and safety issues at IBD diagnosis and during follow-up. Statistical analyses will be performed on clinical parameters such as demography, response to therapy and the main aspect of safety, included in the minimum dataset. Analyses may also be performed on other parameters included all the uploaded datasets.

ELIGIBILITY:
Inclusion Criteria:

* Any patient diagnosed with IBD defined by validated diagnostic criteria can be included into the registry. The criteria for IBD diagnosis were based on previously published criteria for IBD diagnosis, including clinical, endoscopic, laboratory, and histopathological aspects, as well as small bowel imaging studies

Exclusion Criteria:

* Suspected IBD diagnosis without confirmation
* IBD patients with incomplete information about therapy and follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Target population: Any patient diagnosed with IBD defined by validated diagnostic criteria. In order to ensure the inclusion of all IBD patients in Argentina, the executive committee invites all centers associated to GADECCU and involved in the management of IBD patients, regardless of the volume of patients they are in charge of, including both public and private centers. To reduce the possibility of selection bias, each participating physician from each center should aim to include all patients seen in their practice or clinic.
Sampling Method: Non-Probability Sample
Enrollment: 4250 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Demography | Observational from July-2023
  Information from IBD patients in terms of demographic, clinical and diagnostic aspects

SECONDARY OUTCOMES:
Safety aspects of IBD patients | Observational from July-2023
  Safety aspects, including infections, and access to healthcare

OTHER OUTCOMES:
Therapy efectiveness | Observational from July-2023
  For the treatment effectiveness outcome, information about IBD complications as flares, need of hospitalization and surgery will be included

CONTACTS AND LOCATIONS:
Overall Officials: Domingo C Balderramo, MD, PhD, Principal Investigator — Grupo Argentino de Enfermedad de Crohn y Colitis Ulcerosa
Locations (1):
- Hospital Privado Universitario de Cordoba, Córdoba, Córdoba Province, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hracs L, Windsor JW, Gorospe J, Cummings M, Coward S, Buie MJ, Quan J, Goddard Q, Caplan L, Markovinovic A, Williamson T, Abbey Y, Abdullah M, Abreu MT, Ahuja V, Raja Ali RA, Altuwaijri M, Balderramo D, Banerjee R, Benchimol EI, Bernstein CN, Brunet-Mas E, Burisch J, Chong VH, Dotan I, Dutta U, El Ouali S, Forbes A, Forss A, Gearry R, Dao VH, Hartono JL, Hilmi I, Hodges P, Jones GR, Juliao-Banos F, Kaibullayeva J, Kelly P, Kobayashi T, Kotze PG, Lakatos PL, Lees CW, Limsrivilai J, Lo B, Loftus EV Jr, Ludvigsson JF, Mak JWY, Miao Y, Ng KK, Okabayashi S, Olen O, Panaccione R, Paudel MS, Quaresma AB, Rubin DT, Simadibrata M, Sun Y, Suzuki H, Toro M, Turner D, Iade B, Wei SC, Yamamoto-Furusho JK, Yang SK, Ng SC, Kaplan GG; Global IBD Visualization of Epidemiology Studies in the 21st Century (GIVES-21) Research Group. Global evolution of inflammatory bowel disease across epidemiologic stages. Nature. 2025 Jun;642(8067):458-466. doi: 10.1038/s41586-025-08940-0. Epub 2025 Apr 30. PMID 40307548
- [Background] Mak JWY, Sun Y, Limsrivilai J, Abdullah M, Kaibullayeva J, Balderramo D, Vergara BI, Paudel MS, Banerjee R, Hilmi I, Ali RAR, Wei SC, Ng KK, Altuwaijri M, Kelly P, Yamamoto-Furusho JK, Kotze PG, Ahuja V, Chong VH, Dao HV, Abbey Y, Ching JYL, Ho A, Chan AKW, Bernstein CN, Gearry RB, Abreu M, Rubin DT, Dotan I, Hracs L, Kaplan GG, Ng SC; GIVES-21 Consortium. Development of the global inflammatory bowel disease visualization of epidemiology studies in the 21st century (GIVES-21). BMC Med Res Methodol. 2023 May 25;23(1):129. doi: 10.1186/s12874-023-01944-2. PMID 37231405
- [Background] Balderramo D, Quaresma AB, Olivera PA, Savio MC, Villamil MPG, Panaccione R, Ng SC, Kaplan GG, Kotze PG. Challenges in the diagnosis and treatment of inflammatory bowel disease in Latin America. Lancet Gastroenterol Hepatol. 2024 Mar;9(3):263-272. doi: 10.1016/S2468-1253(23)00284-4. PMID 38340754
- [Background] Olivera PA, Balderramo D, Lasa JS, Zubiaurre I, Correa G, Lubrano P, Ruffinengo O, Yantorno M, Rausch A, Pinero G, Bolomo A, Amigo C, El-Hakeh J, Leonardi DB, Brion L, Sambuelli A. Real-world clinical characteristics and therapeutic strategies in patients with moderate-to-severe inflammatory bowel disease in Argentina: Data from the RISE-AR study. Gastroenterol Hepatol. 2025 Oct;48(8):502287. doi: 10.1016/j.gastrohep.2024.502287. Epub 2024 Nov 15. English, Spanish. PMID 39549817
- [Background] Balderramo D, Trakal J, Herrera Najum P, Vivas M, Gonzalez R, Benavidez A, Lopez Villa D, Daino D, Raiden K, German A, Corzo MA, Ponce de Leon J, Ferrer L, German C, Balzola S, Idoeta A, Zarate F, Defago MR; Grupo Cordoba de Cooperacion para el Manejo y Estudio de la Enfermedad Inflamatoria Intestinal (CEMEI Group). High ulcerative colitis and Crohn's disease ratio in a population-based registry from Cordoba, Argentina. Dig Liver Dis. 2021 Jul;53(7):852-857. doi: 10.1016/j.dld.2021.01.006. Epub 2021 Jan 30. PMID 33531211